CLINICAL TRIAL: NCT05236075
Title: Assessment of Tolerance to the Treatment of Obstructive Sleep Apnea by Shear Wave Inducer Collar
Brief Title: Assessment of Tolerance to the Treatment of Obstructive Sleep Apnea by Shear Wave Inducer Collar (ET-SAOS-OC)
Acronym: ET-SAOS-OC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_1339; 2021-A03183-38 (Other: ANSM)
Record Dates: First submitted 2022-01-17; First posted 2022-02-11 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Sleep Apnea
Keywords: obstructive sleep disorders; polysomnography; collar; shear waves
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with polysomnography diagnostic of obstructive sleep disorders moderate to severe (Experimental)
  Interventions: Device: shearing wave collar

INTERVENTIONS:
Device: shearing wave collar — Collar inducing shearing wave to treat obstructive sleep disorders

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common disease, affecting 10-15% of the general adult population. This pathology is characterized by iterative nocturnal episodes of complete or partial obstruction of the upper airways during sleep leading to chronic intermittent nocturnal hypoxia and sleep fragmentation. The number of nocturnal respiratory anomalies per hour of sleep characterizes the severity of the disease with a gradual gradation of severity from mild (from 5 to 15 anomalies per hour) to moderate (15 to 30 anomalies per hour) and severe (over 30 anomalies per hour). The rationale for this severity classification is the increase in morbidity and mortality proportional to the severity of OSA as defined.

OSA is accompanied by a fragmentation of sleep often responsible for excessive daytime sleepiness, causing an increase in occupational accidents with work stoppage and traffic accidents.

The second consequence of repeated nocturnal obstructions is chronic intermittent nocturnal hypoxia which has deleterious cardiovascular effects, constituting an independent cardiovascular risk factor.

Shear waves are elastic waves of low frequency (less than 1000 oscillation per second - 1000Hz). It propagates only in solids and soft solids such as the human body. The propagation of a shear wave generates a reversible micrometric displacement of the particles that make up this medium. The energy of these waves is related to the amplitude of movement of the particles.

Elastography is an imaging modality for measuring the elasticity of biological tissues by shear waves. The shear wave is a mechanical wave sensitive to the change in the elasticity of its propagation medium. This sensitivity is manifested by the variation of its propagation speed. Hardness results in acceleration of the wave and softness in its slowing down.

The therapeutic use of shear waves has never been used for the treatment of sleep apnea but its use could be an additional therapeutic arsenal of Continuous Positive Pressure.

The technology developed by BREAS MEDICAL AB is based on the use of shear waves for the treatment of sleep apnea. The treatment is delivered using a cervical collar equipped with six sources (vibrating pistons) generating shear waves. The treatment generates shear waves at frequencies that vary from 20 to 250 Hz continuously, and at amplitudes less than 50 microns of the same order of magnitude of vibration as snoring. In view of the innovative nature of the treatment, the medico-technical team of BREAS MEDICAL AB carried out an analysis of the risks related to the device and to the propagation of waves, including the norms and standards imposed by the competent bodies.

The investigators would like, in a first-dose study in humans, to assess safety in patients with sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* aged 30 to 69 in order to avoid tissue changes in the older age groups of the adult population
* patients with polysomnography diagnosic of obstructive sleep disorders moderate to severe
* referred to the Sleep Center of the Croix Rousse Hospital for sleep disorders and suspected of having a sleep apnea syndrome when first making contact in consultation or by phone call.
* All patients accepting the additional 24 hours instead of the usual 24 hours, ECG, neck vessel Doppler and trial shear wave therapy. This second night will be scheduled at the end of the first night.
* Patients agreeing to spend this second night in a period of less than 15 days between the first night and the second night
* Patient without fever >38°C
* having communicated their signed consent
* Affiliated with a social security scheme
* Having a negative PCR covid test in the last 48 hours prior to hospitalization, if used during the protocol.

Exclusion Criteria:

* Patient with a cardiac pace maker
* Patient with a tracheostomy
* Patient with cancerous disease during treatment
* Persons referred to in articles L1121-5 to L1121-8 of the CSP (pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure, cannot be included in clinical trials
* Patient unable to remove their dentures if concerned
* Patients with vascular plaques seen on cervical Doppler
* Patient having presented a pathology in the previous months which contraindicates the continuation of the study at the discretion of one of the medical investigators (new cardiac pathology of less than 3 months, or of 6 months and not stabilized, vascular accident cerebral or transient ischemic attack of less than 3 months, other pathologies of less than 3 months at the discretion of the investigator).
* Patients with any known cutaneous or deep cervical abnormality (dermatosis, glottic abnormality, Zencker's diverticulum, Basedow, toxic thyroid nodule(s), parathyroid adenoma or hyperplasia, wound, recent scar, burn, etc.)
* Patients with an implanted electronic device, medical or not; other than implanted automatic pacemakers or pacemakers and defibrillators (cochlear implant, brain implants, RFID chip).
* Patients suffering from Central nervous sytem disorder such as epilepsy, Parkinson disease.
* Patients with a cervical malformation or a particular cervical morphology (very wide neck outside collar size range, goiter, etc.) incompatible with the characteristics of the collar.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
feasibility of wearing the shear wave collar | Day after the polysomnographic night (Day1 or Day15)
  The feasibility of wearing the shear wave collar will be determined by the percentage of patients who have worn the collar at least 60% of their night AND who agree to wear this shear wave diffuser collar again if treatment is necessary.
  The duration collar wearing will be the delay in minutes between the putting on of the collar by a nurse and the removal of the collar by the patient or a nurse. The night duration will be the total duration of sleep in minutes determined by the polysomnography measures. The exact times (accuracy in second) of putting on and taking off the collar will be collected via the collar sensors specifically provided for this purpose. After each session, collar data are extracted by the BREAS technician and entered into the patient medical file and the eCRF.

SECONDARY OUTCOMES:
Sleep quality | Day after the polysomnographic night (Day1 or Day15)
  quality of sleep according to the patient will be assessed using the question: "I am satisfied with my night" with a 5-level Likert scale: very satisfied, satisfied, no opinion, moderately satisfied, not satisfied
confort during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "How do you judge the collar confort" with a 5-level Likert scale: very satisfied, satisfied, no opinion, moderately satisfied, not satisfied
vibration occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "How do you judge the collar vibration" with a 5-level Likert scale: very satisfied, satisfied, no opinion, moderately satisfied, not satisfied
Noise occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "How do you judge the collar noise" with a 5-level Likert scale: very satisfied, satisfied, no opinion, moderately satisfied, not satisfied
inconveniences due to the collar lock | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "How do you judge the collar lock" with a 5-level Likert scale: very satisfied, satisfied, no opinion, moderately satisfied, not satisfied
redness occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "Do you have redness" with a 4-level Likert scale: None, Light, moderate, intense
Burnt occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "Do you have Burnt " with a 4-level Likert scale: None, Light, moderate, intense
blisters occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  inconveniences according to the patient will be assessed using the question: "Do you have blisters " with a 4-level Likert scale: None, Light, moderate, intense
Pain occurring during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  Pain according to the patient will be assessed using the question using anumeric scale from 0 to 10, 0 being the absence of pain and 10 the worst pain experienced
Hypertension safety | Day after the polysomnographic night (Day1 or Day15)
  Hypertension evolution between before and 1 day after the polysomnographic night will be measures in mmHg
cardiac frequency safety | Day after the polysomnographic night (Day1 or Day15)
  cardiac frequency evolution between before and Day after the polysomnographic night will be measures in mean frequency
adverse event post evaluation | 7 Days after the second polysomnographic night (Day8 or Day22)
  Adverse event related to the night wearing the collar declared in the 7 days following the second polysomnographic night.
Sleep Apnea severity during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  Sleep Apnea severity will be evaluated with the apnea-hypopnea index
Sleep fragmentation during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  Sleep fragmentation level will be evaluated with the number of micro wake-up
duration of sleep stage during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  duration of sleep stage in minutes
sleep efficacy during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  sleep efficacy will be measured using the index time of real sleep in minutes divided by the time spent in bed in minutes
Night oxygen saturation during the night wearing the collar | Day after the polysomnographic night (Day1 or Day15)
  Night oxygen saturation will be measured using the SaO2 mean

CONTACTS AND LOCATIONS:
Locations (1):
- Department of sleep and respiratory disorders, Hopital Nord Croix-Rousse - Hospices Civils de Lyon, Lyon, France